CLINICAL TRIAL: NCT05329090
Title: Evaluation of Glucocorticoids Plus Rituximab Compared to Glucocorticoids Plus Placebo for the Treatment of Patients with Newly-Diagnosed or Relapsing IgA Vasculitis: a Prospective, Randomized, Controlled, Double-blind Study
Brief Title: Evaluation of Glucocorticoids Plus Rituximab in Patients with Newly-Diagnosed or Relapsing IgA Vasculitis
Acronym: RIGA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hopital Foch (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019_0068
Record Dates: First submitted 2021-08-09; First posted 2022-04-14 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: IgA Vasculitis
Keywords: Rituximab
MeSH Terms: conditions — IgA Vasculitis | interventions — Rituximab

STUDY DESIGN:
Intervention Model Description: Design of trial :
  * Controlled (the comparator is a Placebo)
  * Randomised
  * Double blind
  * Parallel groupe
  * With a double layering
Who Masked: Participant, Investigator
Masking Description: This trial will be comparative, randomized, double-blind and double-dummy in order to limit performance and evaluation bias.
  Neither patients, nor physicians will know the treatments allocated to their patients.
  Investigators will be in blind of the leukocyte formula during all study period, from day 1.
  Neither patients, nor physicians will know the treatments allocated to their patients.
  Investigators will be in blind of the CD19+ count during all study period, from day 15.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental group (Experimental): Experimental therapeutic strategy based on the use of rituximab in combination with glucocorticoids
  Interventions: Drug: Rituximab Injection
- control group (Placebo Comparator): Control therapeutic strategy based on glucocorticoids plus placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Rituximab Injection — anti-CD20 monoclonal antibody leading to B-cell depletion, in relapsing and/or refractory IgAV patients
  Other Names: Rixathon; Truxima
  Arms: experimental group
Drug: placebo — placebo experimental treatment
  Other Names: NaCl
  Arms: control group

SUMMARY:
Systemic vasculitis are inflammatory diseases of the blood vessels, responsible for systemic manifestations. Among the systemic vasculitis affecting small blood vessels, IgA vasculitis (IgAV) is one of the most common forms and mainly affects the skin, joints, kidneys and gastrointestinal tract. Kidney and gastrointestinal damage can be serious, causing complications and life-threatening sequelae, especially in adults. The treatment of adult-onset IgAV is still a matter of debate. Glucocorticoids have been the standard of care for inducing remission for years in severe forms of IgAV. However, not all patients achieve remission and may experience disease flares associated with increased morbidity and mortality. In addition, the cumulative side effects of glucocorticoids are also major causes of long-term adverse events and death.Rituximab (RTX), an anti-CD20 monoclonal antibody, has been shown to be spectacularly effective in inducing remission in d 'other small vascular vessels, in particular ANCA-associated vasculitis and cryoglobulinemic vasculitis, with an acceptable safety profile.

Recently, a multicenter observational study suggested that RTX was an effective and safe therapeutic option for treating relapsed and / or refractory adult IgAV.

Overall, RTX may be an effective and safe therapeutic approach in adult IgAVs, justifying the need for a prospective randomized controlled trial evaluating Rituximab as an induction of remission for adult IgAV.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven diagnosis of IgAV according to Chapel Hill Consensus Conference definitions
* Patient aged of 18 years or older
* Patients with newly-diagnosed disease or relapsing disease at the time of screening, with an active disease defined by active manifestations attributable to IgAV
* Patients with severe involvement of at least one organ
* Patients within the first 21 days following initiation/increase of glucocorticoids at a dose < 1 mg/kg/day
* Has signed an informed consent form prior to any study related procedures
* Affiliated to a national health insurance

Exclusion Criteria:

* Patients with ANCA-associated vasculitis, or other vasculitis, defined by the ACR criteria and/or the Chapel Hill Consensus Conference,
* Patients with IgAV in remission of the disease,
* Patients with severe cardiac failure defined as class IV in New York Heart Association,
* Patients with severe, uncontrolled cardiac disease,
* Patients with acute infections or chronic active infections (including HIV, HBV or HCV),
* Patients with active cancer or recent malignancy (<5 years), except basocellular carcinoma and prostatic cancer of low activity controlled by hormonal treatment,
* Pregnant women and breastfeeding. Patients with childbearing potential must use reliable contraceptive methods throughout the study and at least for 12 months after the last study drug administration,
* Patients with IgAV who have already been treated with rituximab within the previous 12 months,
* Patients treated with immunosuppressive therapy within the last 3 months,
* Patients with hypersensitivity to human or chimeric monoclonal antibodies,
* Patients with contraindication to use rituximab,
* Patients treated with any concomitant drugs contraindicated for use with the rituximab according to its SmPC,
* Patients with contraindication to use routine care treatments (Glucocorticoids, Angiotensin-converting-enzyme (ACEis) or angiotensin receptor blockers (ARBs), dexchlorphéniramine),
* Patients in a severely immunocompromised state,
* Patients with other uncontrolled diseases, including drug or alcohol abuse, severe psychiatric disorders, that could interfere with his/her compliance to protocol requirements,
* Patients currently participating in another clinical study or 3 months prior to randomization,
* Patients suspected not to be observant to the proposed treatments,
* Patients unable to give written informed consent prior to participation in the study
* Being deprived of liberty or under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2025-07-16 (Estimated); Study Completion 2026-01-16 (Estimated)

PRIMARY OUTCOMES:
Rituximab efficacy | 180 days
  The proportion of patients alive who achieved remission with a prednisone dose of 0 mg/day at 180 days
Rituximab efficacy | 360 days
  The proportion of patients alive who achieved remission with a prednisone dose of 0 mg/day at 360 days

SECONDARY OUTCOMES:
Efficacy of rituximab-based regimen to induce remission | 180 days
  Proportion of patients with BVAS=0 (or BVAS of ≤5 if all scores were due to persistent hematuria or proteinuria) and a prednisone dose ≤5 mg/day at 180 days
Efficacy of rituximab-based regimen to induce remission | 360 days
  Proportion of patients with BVAS=0 (or BVAS of ≤5 if all scores were due to persistent hematuria or proteinuria) and a prednisone dose ≤5 mg/day at 360 days
Assessement the duration of remission | 360 days
  Proportion of patients achieving remission for ≥3 consecutive months over the 360 days, with BVAS=0 (or BVAS of ≤5 if all scores were due to persistent hematuria or proteinuria) and a prednisone dose ≤5 mg/day at 360 days.
Assessment of patients achieving a complete or partial renal remission & renal outcome remission | 180 days
  Proportion of patients in complete renal and partial renal remission at 180 days (Renal parameters at 180 days compared with baseline: eGFR, daily proteinuria, hematuria, arterial hypertension, use of angiotensin converting enzyme inhibitor, occurrence of end-stage renal disease)
Assessment of patients achieving a complete or partial renal remission & renal outcome remission | 360 days
  Proportion of patients in complete renal and partial renal remission at 360 days (Renal parameters at 360 days compared with baseline: eGFR, daily proteinuria, hematuria, arterial hypertension, use of angiotensin converting enzyme inhibitor, occurrence of end-stage renal disease)
Measure of glucocorticoids dose | 160 days
  Area under the curve for prednisone dose at 180 days in the two treatment groups
Measure of glucocorticoids dose | 360 days
  Area under the curve for prednisone dose at 360 days in the two treatment groups
Number of participants with adverse events for the safety analyse | 360 days
  Adverse events, expressed as adverse events according to the CTCAE toxicity grading system per patient-year at days 180 and 360 for the following adverse events combined: death (all causes), grade 2 or higher leukopenia or thrombocytopenia, grade 3 or higher infections, malignancies, venous thromboembolic events, hospitalization resulting either from the disease or from a complication due to the study treatment, infusion reactions (within 24 hours of infusion) that result in the cessation of further infusions, death
The sequelae assessed by the Vasculitis Damage Index | 180 days
  The Vasculitis Damage Index in the two treatment groups
The sequelae assessed by the Vasculitis Damage Index | 360 days
  The Vasculitis Damage Index in the two treatment groups
Quality of life of patients | 180 days
  HAQ and SF-36 questionnaires at 180 days
Quality of life of patients | 360 days
  HAQ and SF-36 questionnaires at 360 days
Patient reported outcome | 360 days
  The patient-reported outcomes (PRO) including patient-reported disease activity, anxiety and depression, burden of the disease and treatment and adherence to treatment, at days 180 and 360 after randomization in the two treatment groups, and during the long-term follow-up
Patient survival | 360 days
  Number of patient survival

CONTACTS AND LOCATIONS:
Overall Officials: Romain Paule, Dr, Principal Investigator — Hôpital Foch
Locations (13):
- France (13):
  - Hopital La Cavale Blanche, Brest
  - CHU Clermont Ferrand, Clermont-Ferrand
  - Hôpital Edouard Herriot, Lyon
  - CHU Marseille, Marseille
  - APHM de La Timone, Marseille
  - Hôpital André Grégoire, Montreuil
  - CHU Nantes, Nantes
  - CHU Nîmes (Caremeau), Nîmes
  - Hôpital Cochin, Paris
  - CHU Strasbourg, Strasbourg
  - Hôpital Foch, Suresnes
  - CHU Toulouse, Toulouse
  - CHRU Bretonneau, Tours

IPD SHARING:
Plan to Share IPD: No